CLINICAL TRIAL: NCT01823120
Title: Text Message Intervention to Reduce Repeat Self-harm in Patients Presenting to the Emergency Department
Brief Title: Text Message Intervention to Reduce Repeat Self-harm
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resignation of critical volunteer staff and lack of funding
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Beaumont Hospital (Other); Royal College of Surgeons, Ireland (Other)
Responsible Party: Principal Investigator, Vincent Agyapong, Dr, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13/18
Record Dates: First submitted 2013-03-26; First posted 2013-04-04 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Self-Injurious Behavior
Keywords: Self harm; Emergency Department; Repetition; Supportive Text messages; Interactive
MeSH Terms: conditions — Self-Injurious Behavior; Emergencies | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No text messages (No Intervention): Patients in the non-intervention group will not receive any text messages. However, they will also receive the routine outpatient follow-up arrangements associated with attendance at an ED with self-harm including the provision of a contact phone number for the Samaritans.
- Supportive and interactive text messages (Experimental): We will deliver daily supportive and informative text messages for one month followed by one supportive and informative text message every other day the second month and then one weekly text message the third month to patients in the intervention group after they have been discharged from the ED following an episode of self-harm. Supportive text messages will mainly target relieving the patients of mood symptoms and providing them with strategies for dealing with suicidal thoughts while the informative ones will provide patients with a dedicated mobile phone number through which they can receive interactive support from the Samaritans. The text messages will encourage participants to text the Samaritans in times of crisis. Please see appendix I for examples of the relevant text messages.
  Interventions: Other: Supportive and interactive text messages

INTERVENTIONS:
Other: Supportive and interactive text messages
  Arms: Supportive and interactive text messages

SUMMARY:
Between 6% and 30% of people who harm themselves repeat this self-harm within the following 12 months. The investigators know that people who harm themselves are much more likely to commit suicide, but the investigators have no clear evidence about the best way to reduce the likelihood of someone harming themselves again.

Text messaging is now a common form of communication. Previous research has shown us that the investigators can use text messages for different types of health care interventions. Examples of this include reminding patients of medical appointments, delivering test results, to check patient side effects following treatment and to reduce depressive symptoms in patients with depression and alcohol problems. The Samaritans have introduced interactive text messages (where you can have a conversation by text with their service) and have noted an increasing use of this contact with their service.

This research study is taking place to find out if using supportive and interactive text messages can reduce further episodes of self-harm in patients who present to the Emergency Department (ED) with self-harm.

The investigators hypothesize that supportive, informative and interactive text messages delivered to patients discharged from an ED after an episode of self-harm will significantly reduce the frequency and intensity of thoughts of self-harm and self-harming behaviour in patients compared with those receiving only follow-up treatment as usual. A secondary hypothesis is that patients receiving the text messages will report a favourable experience and an overall satisfaction with the system.

DETAILED DESCRIPTION:
Repetition of self-harm is common, ranging from 6% to 30% in 12 months. Repetition is strongly associated with subsequent suicide and has important implications for healthcare resources. In every country including Ireland, fatal suicide attempts rank among the top ten causes of death for individual of all ages and one of the three leading causes of death in the 15 -35 years age group.

Previous studies of interventions to reduce the repetition of self-harm in unselected patient groups have been unsuccessful in reducing the proportion of repeaters. These interventions have included the use of antidepressants, problem solving, intensive care with outreach, an emergency card, psychosocial crisis intervention, and guaranteed inpatient shelter in cases of emergency. In a study involving the use of low cost postcards after an episode of self-poisoning, although no significant difference in the proportion of individual patients who repeated self-harm were detected, there was a clinically and statistically significant reduction in the number of events per individual by about 50%.

Only a few non-pharmacological interventions have been reported to be effective in reducing repetition in selected subsets of populations with self-harm including; partial hospitalization, dialectical behaviour therapy and psychodynamic interpersonal therapy. These interventions are all resource intensive and therefore may only be applicable to carefully selected patients.

Given the recent global financial crisis with consequent diminution of health care resources, interventions are needed that could be delivered economically to entire populations of patients who self-harm. In light of the growing interest in using text messages as an intervention in healthcare, the investigators will focus in this study on exploring the potential for using text messages to reduce repeat self-harm in patients presenting to the Emergency Department (ED).

There is established research evidence for using text messages to remind patients of scheduled medical appointments, to coordinate medical staff,to deliver medical test results and to monitor patient side effects following treatment.

In a review of the literature on the use of text messaging for clinical and healthy behaviour interventions, Wei et al. (2011) found that among 16 randomized controlled trials, 10 reported significant improvement with interventions and six reported differences suggesting positive trends. In one meta-analysis of four randomised trials of mobile phone-based interventions for smoking cessation, it was reported that text message interventions resulted in a significant increase in short-term self-reported quitting (RR of 2.18, 95% CI 1.80 to 2.65). In the same review, when data from an internet and a mobile phone programme were pooled and meta-analysed, they found significant increases in both short-, and long-term, self-reported quitting (RR of 2.03, 95% Conficence Intervals (CI)= 1.40 to 2.94).

In a study of text message services based on qualitative interviews with 12 young people, the aim of which was to provide young people with information on cannabis and help them to reduce their consumption of the drug, participants reported that they saw the messages as flexible and discrete, and as being personally meant for them. They paid more attention to the messages than they did to mass approaches such as public information broadcasts on TV. Along with other factors, the participants reported feeling motivated to decrease their level of cannabis abuse and to maintain a reduced level. .

In another study, young adults in 3 urban EDs (n= 45; aged 18 to 24 years, 54% women) who were identified as hazardous drinkers by the Alcohol Use Disorders Identification Test-Consumption Score were randomly assigned by the researchers to weekly text message-based feedback with goal setting (Intervention), weekly text message-based drinking assessments without feedback (Assessment), or to a control who received no text messages. At 3 months, they found that participants who were exposed to the text message-based intervention had 3.4 (Standard Deviation (SD)= 5.4) fewer heavy drinking days in the last month and 2.1 (SD 1.5) fewer drinks per drinking day when compared to baseline.

In a recent randomised trial in Ireland of supportive text messages for patients with depression and comorbid alcohol use disorder, there was a trend towards finding a greater cumulative abstinence duration in the group that received twice daily supportive text messages compared to the control group who only received fortnightly tank you text messages: 88.3 (SD=6.2) vs. 79.3 (SD=24.1), t=1.78, df=48, p=0.08. In this trial, after adjusting for baseline scores, patients in the supportive text message group also had significantly lower Beck's Depression Inventory Scores compared to the control groups; 8.5 (SD=8.0) vs. 16.7 (SD=10.3) respectively, F (1, 49) = 9.54, p=0.003, ƞp2=0.17.

In a study by Owens et al. (2010) to engage a group of self-harmers in the development of a text-messaging intervention to reduce repetition of self-harm, three broad categories of message emerged, namely, those that affirmed or validated emotions (e.g. "it's ok to feel angry"), those that prescribed actions, distractions or cognitive strategies (e.g. "call Samaritans," "have a warm bath"," take it a minute at a time") and those that were interrogative or designed to initiate dialogue (e.g. "do you want to talk?"). They also found that the group were unable to reach an agreement on a set of messages that might work in all circumstances to reduce the urge to self-harm or to enable people to feel cared for, concluding instead that text messages may need to be individualised. A major limitation of this study was its small sample size of only 8 people. Furthermore, participants in this study only reported how they envisaged they would respond to text messages rather than how they actually responded to text messages which could vary significantly from what is reported. In the recent randomised trial in Ireland of generic supportive text messages for patients with depression and comorbid alcohol use disorder, 20 of the 24 patients (83%) reported that the intervention had played a useful role in helping to improve their mental health.

Recently, the Samaritans in Ireland introduce a limited interactive text message programme for patients who experience suicidal ideation. This service allows clients to receive support when in crisis via an interactive text messaging programme from a trained volunteer.

After an extensive review of the literature using Google Scholar, MEDLINE, Pub Med, ERIC, Web of Science, Science Direct and PsychINFO, no published randomised trial was found on the use of text messages delivered via mobile phone as an intervention to address suicidal ideation and repeat self-harm in patients presenting with self-harm to the ED. Thus, the investigators seek to determine if text messaging is a useful and effective strategy to help reduce the frequency and intensity of thoughts of self-harm and depressive symptoms after patients are discharged from an ED following a presentation with self-harm.

The investigators hypothesize that supportive, informative and interactive text messages delivered to patients discharged from an ED after an episode of self-harm will significantly reduce the frequency and intensity of thoughts of self-harm and self-harming behaviour in patients compared with those receiving only follow-up treatment as usual. A secondary hypothesis is that patients receiving the text messages will report a favourable experience and an overall satisfaction with the system.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years and over, presenting to the ED with self-harm.
* All patients should have a mobile phone, be familiar with text messaging technology and be willing to take part in the study.

Exclusion Criteria:

* Patients who do not consent to take part in the study.
* Patients who do not have a mobile phone or are unable to use the mobile text message technology.
* Patients who are admitted as a psychiatric inpatient following the assessment in the ED or those who require admission to a medical ward for longer than 48 hours.
* Patients who would be unavailable for follow-up during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Repetition of self-harm | Three months
  Proportion of patients repeating self-harm
Change scores on the Suicide Behaviors Questionnaire from baseline | Baseline and three months
  The change scores on the Suicide Behaviors Questionnaire from baseline

SECONDARY OUTCOMES:
Repeat episodes of self-harm per person | Three months
  Number of repeat episodes of self-harm per person
Change scores in the Modified Scale for Suicide Ideation from baseline | Baseline anf three months
  The change scores on the Modified Scale for Suicide Ideation from baseline
Change scores on the Positive and Negative Suicide Ideation Inventory from baseline | Baseline and three months
  The change scores on the Positive and Negative Suicide Ideation Inventory from baseline
Change scores on the Beck Hopelessness Scale from baseline | Baseline and three months
  The change scores on the Beck Hopelessness Scale from baseline
Change scores on the Global Assessment of Functioning Scale from baseline | Baseline and three months
  The change scores on the Global Assessment of Functioning Scale from baseline

OTHER OUTCOMES:
Utilisation of the services provided by the Samaritans Ireland | Three months
  The range and frequency of utilisation of the services provided by the Samaritans Ireland
Patient satisfaction with treatment | Three months
  Patient satisfaction (for both groups) with their overall follow-up treatment at three months following discharge from the ED would be measured using a self-designed likert scale.
Feedback about patients' experiences, expectations and satisfaction with the communication system | Three months
  Feedback about patients' experiences, expectations and satisfaction with the communication system and its perceived impact on their mood, suicidal thoughts and potential to repeat self-harm. These aspects would be measured using semi-structured questionnaires which include likert scales at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Vincent IO Agyapong, MRCPsych MD, Principal Investigator — University of Dublin, Trinity College Dublin; Siobhan MacHale, FRCPsych, Study Chair — Beaumont Hospital Dublin
Locations (1):
- Beaumont Hospital, Dublin, Co Dublin, Ireland

REFERENCES:
- [Background] Agyapong, V., J. Milnes, M. McLoughlin and C. Farren (2012).
- [Background] Agyapong, V. I. O., M. D. McLoughlin and C. K. Farren. Usefulness of Supportive Text Messages to Patients with Alcohol Use Disorder and Comorbid Depression-A Single-Blind Randomised Controlled Trial. J. Affect. Disord. Volume 141, Issues 2-3, 10 December 2012, Pages 168-176
- [Background] Australian Bureau of Statistics (2003). Household Use of Information Technology Canberra, Australia. B., P. (2003).
- [Background] Bateman, A. and P. Fonagy (1999).
- [Background] Brianna S., Fjeldsoe B.A. and Alison L. (2009).
- [Background] Carter, G. L., K. Clover, I. M. Whyte, A. H. Dawson and C. D'Este (2005).
- [Background] Cohen, J. (1988). Statistical power analysis for the behavioral sciences, Academic Press. New York. Downer, S., J. Meara and A. Da Costa (2005).
- [Background] Guthrie E, Kapur N, Mackway-Jones K, Chew-Graham C, Moorey J, Mendel E, Marino-Francis F, Sanderson S, Turpin C, Boddy G, Tomenson B. Randomised controlled trial of brief psychological intervention after deliberate self poisoning. BMJ. 2001 Jul 21;323(7305):135-8. doi: 10.1136/bmj.323.7305.135. PMID 11463679
- [Background] Hawton K, Arensman E, Townsend E, Bremner S, Feldman E, Goldney R, Gunnell D, Hazell P, van Heeringen K, House A, Owens D, Sakinofsky I, Traskman-Bendz L. Deliberate self harm: systematic review of efficacy of psychosocial and pharmacological treatments in preventing repetition. BMJ. 1998 Aug 15;317(7156):441-7. doi: 10.1136/bmj.317.7156.441. PMID 9703526
- [Background] Haynes RB., S. D., Guyatt G., Tugwell, P., (2005). Clinical Epidemiology: How to do Clinical Practice Research. Philadelphia PA, Lippincott, Williams, Wilkins.
- [Background] House A, Owens D, Patchett L. Deliberate self harm. Qual Health Care. 1999 Jun;8(2):137-43. doi: 10.1136/qshc.8.2.137. No abstract available. PMID 10557677
- [Background] Jeffery RW, Drewnowski A, Epstein LH, Stunkard AJ, Wilson GT, Wing RR, Hill DR. Long-term maintenance of weight loss: current status. Health Psychol. 2000 Jan;19(1S):5-16. doi: 10.1037/0278-6133.19.suppl1.5. PMID 10709944
- [Background] Leong KC, Chen WS, Leong KW, Mastura I, Mimi O, Sheikh MA, Zailinawati AH, Ng CJ, Phua KL, Teng CL. The use of text messaging to improve attendance in primary care: a randomized controlled trial. Fam Pract. 2006 Dec;23(6):699-705. doi: 10.1093/fampra/cml044. Epub 2006 Aug 17. PMID 16916871
- [Background] Linehan MM, Armstrong HE, Suarez A, Allmon D, Heard HL. Cognitive-behavioral treatment of chronically parasuicidal borderline patients. Arch Gen Psychiatry. 1991 Dec;48(12):1060-4. doi: 10.1001/archpsyc.1991.01810360024003. PMID 1845222
- [Background] Luborsky, L. (1962).
- [Background] Menon-Johansson AS, McNaught F, Mandalia S, Sullivan AK. Texting decreases the time to treatment for genital Chlamydia trachomatis infection. Sex Transm Infect. 2006 Feb;82(1):49-51. doi: 10.1136/sti.2004.014381. PMID 16461603
- [Background] Molenberghs G, K. M., Ed. (2007). Missing data in clinical studies. Chichester, John Wiley & Sons. Owens, C., P. Farrand, R. Darvill, T. Emmens, E. Hewis and P. Aitken (2011).
- [Background] Patrick K, Raab F, Adams MA, Dillon L, Zabinski M, Rock CL, Griswold WG, Norman GJ. A text message-based intervention for weight loss: randomized controlled trial. J Med Internet Res. 2009 Jan 13;11(1):e1. doi: 10.2196/jmir.1100. PMID 19141433
- [Background] Rice R. and K. J. (2003).
- [Background] Rickards L., Fox K., Roberts C., Flectcher L. and G. E. (2004). Living in Britain-The 2002 General Household Survey. London: Office for National Statistics. London, Office for National Statistics.
- [Background] Sherry E, C. B., Warnke P. (2002).
- [Background] Stross, R. (2008). What carriers aren't eager to tell you about texting. New York Times. New York.
- [Background] Tomnay JE, P. M., Fairley CK. (2005).
- [Background] van der Sande R, Buskens E, Allart E, van der Graaf Y, van Engeland H. Psychosocial intervention following suicide attempt: a systematic review of treatment interventions. Acta Psychiatr Scand. 1997 Jul;96(1):43-50. doi: 10.1111/j.1600-0447.1997.tb09903.x. PMID 9259223
- [Background] Weaver A, Young AM, Rowntree J, Townsend N, Pearson S, Smith J, Gibson O, Cobern W, Larsen M, Tarassenko L. Application of mobile phone technology for managing chemotherapy-associated side-effects. Ann Oncol. 2007 Nov;18(11):1887-92. doi: 10.1093/annonc/mdm354. Epub 2007 Oct 5. PMID 17921245
- [Background] Wei, J., I. Hollin and S. Kachnowski (2011).
- [Background] Whittaker, R., R. Borland, C. Bullen, R. Lin, H. McRobbie and A. Rodgers (2009).
- [Background] Suffoletto , B., C. Callaway, J. Kristan, K. Kraemer and D. B. Clark (2011 Dec 14).
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793